CLINICAL TRIAL: NCT06559839
Title: Vestibular Innovation in Pain: An Open Label Trial
Brief Title: Vestibular Innovation in Pain
Acronym: VIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Michael H Kaplan, Assistant Professor of Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-23-00885
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Pain; Fatigue; Quality of Life
MeSH Terms: conditions — Pain; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fibromyalgia (Experimental): Patients in this arm meet ACR 2011 criteria for Fibromyalgia.
  Interventions: Other: Vestibulocortical Stimulation
- Myalgic Encephalomyelitis/Chronic Fatigue Syndrome, Long Covid, Post Treatment Lyme Disease Syndrome (Experimental): Participants in this arm meet criteria for at least one of the following diseases: Myalgic-Encephalomyelitis/chronic fatigue syndrome (ME/CFS), Long COVID, or Post Treatment Lyme Disease Syndrome.
  Interventions: Other: Vestibulocortical Stimulation

INTERVENTIONS:
Other: Vestibulocortical Stimulation — 50cc of cold water (4℃) irrigated to the right external ear canal, at 1-2 cc/second, with the patient laying supine.
  Other Names: VCS

SUMMARY:
The VIP trial will assess the effectiveness, tolerability, and durability of effect of vestibulocortical stimulation (VCS) - a safe & cost-effective bedside technique - in treating pain, fatigue & related symptoms using validated patient-reported outcomes. Data from this trial will be used to guide optimized treatment protocols in future randomized controlled trials and help inform the implementation of VCS into standard clinical practice.

DETAILED DESCRIPTION:
VCS is a form of non-invasive neuromodulation whereby cold water is irrigated into the external ear canal.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Age equal to or >18 years old
* Stated interest in and willingness to receive VCS and to complete the online patient reported outcomes before and after the procedure.
* Owns or has access to a smart phone or computer to complete outcome measures
* Diagnosis of one of the following:

  * Fibromyalgia (FM), with at least a 4/10 average baseline pain on the numeric rating scale at the time of inclusion.
  * Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS)
  * Long-COVID
  * Post Treatment Lyme Disease Syndrome (PTLDS)

Exclusion Criteria:

An individual with any of the following criteria will be excluded from participation in this study:

* History of tympanic membrane injury, rupture, or surgery

  * Including tympanostomy, or "ear tubes," and/or cochlear implant.
* Ear infection within the last 3 months, or current ear pain.
* Current pregnancy
* Bipolar Disorder
* History of seizures (including non-epileptiform seizures)
* History of syncope
* Inability to lay supine for 30 minutes
* Clinically significant medical, psychological, or behavioral conditions that, in the opinion of the investigator, would compromise participation in the study
* Not fluent in English
* History of or current Meniere's Disease
* History of myocardial infarction (MI), stroke or TIA, or coronary artery bypass graft (CABG) in the last three months
* History of hospitalization for severe hypertension
* History of vestibular schwannoma or meningioma resection.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Change in Diary pain numeric rating scale (Pain NRS) scores | Baseline and at 1 week after VCS
  Change in diary pain scores on a 11 point numeric rating scale at 1 week after VCS as compared to baseline. Full scale from 0-10, with higher score indicating worse pain.

SECONDARY OUTCOMES:
Acute and Longitudinal Change in numeric rating scale (Pain NRS) | Baseline and at 30 minutes, 24 hours, 2 weeks, and 4 weeks
  Pain scores on an 11 point numeric rating scale at 30 minutes, 2 weeks, and 4 weeks after VCS as compared to baseline. Full scale from 0-10, with higher score indicating worse pain.
Percentage of Patients with Numeric Rating Scale (NRS) pain scores > = to 30% and 50% | 30 minutes, 24 hours, 1 week, 2 weeks, 4 weeks
  Percentage of patients with change in pain assessed by NRS pain scores > equal to 30% and 50%. NRS full scale from 0-10, with higher score indicating worse pain.
Brief Pain Inventory- Short Form | 24 hours
  A 9-item instrument. Question 2 which is a diagram and question 7 which asks about medications, will be excluded. Total score from 0 to 10, with higher score indicating worse outcomes.
Patient-Reported Outcomes Measurement Information System (PROMIS-29) Score | 1 week, 2 weeks, 4 weeks
  Patient-Reported Outcomes Measurement Information System 29 (PROMIS-29) measures seven domains: depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and the ability to participate in social roles and activities. Each domain has 4 questions ranked on a 5-point scale, and refer to the 7 previous days except physical function which has not time frame.
  Scoring is standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points.
  Higher scores indicate poorer health outcomes for anxiety, depression, fatigue, ability to participate in social roles and activities, and pain interference domains.
  Lower scores reflect worse outcomes for physical function and sleep disturbances domains.
Overall Well Being Numeric Rating Scale (NRS) | at 30 minutes
  Overall well-being scores on an 11 point numeric rating scale at 30 minutes. NRS full scale from 0-10, with higher score suggesting greater overall wellbeing.
VCS Tolerability Survey | 24 hours post VCS
  A seventeen question tolerability instrument developed specifically for caloric stimulation to assess tolerability by measuring the frequency and intensity of headaches, nausea, and vertigo. The tolerability scale does not have a total score just individual questions re headache nausea vertigo discomfort and grades intensities rated on a 0-10 scale, higher numbers reflecting higher severity of symptoms.
Patient Global Impression of Change (PGIC) Score | 24 hours, 1 week, 2 week, 4 weeks
  The Patient's Global Impression of Change (PGIC) will be used to assess pain. It will evaluate pain from no change (score 0-1), minimally improved (score 2-3), much improved (score 4-5), and very much improved (score 6-7). The patients will answer the following question: "Since beginning treatment at this program, how would you describe the change (if any) in activity limitations, symptoms, emotions, and overall quality of life related to your condition?". Full score from 0-7, with higher score indicating more improvement.
Fatigue Severity Scale (FSS) Score | 1 weeks, 2 weeks, 4 weeks
  A 9-item scale, each item scored from 1 (strongly disagree) to 7 (strongly agree). Total scale from 9-63, with higher score indicating greater fatigue.
Epworth Sleepiness Scale (ESS) Score | 1 weeks, 2 weeks, 4 weeks
  The Epworth Sleepiness Scale (ESS) is an 8-item measure that asks about the probability of dozing or sleeping during typical daytime activities. Scores correlate well with objective measures of speed of daytime sleep onset. The test is a list of eight situations in which the participate rates tendency to become sleepy on a scale of 0, no chance of dozing, to 3, high chance of dozing for each item. Total scale from 0 to 24, with higher score indicating severe excessive daytime sleepiness.
Compass-31 Score | 1 weeks, 2 weeks, 4 weeks
  The COMPASS-31 (Composite Autonomic Symptom Score) is a comprehensive questionnaire used to evaluate symptoms of autonomic dysfunction in various body systems. It contains 31 questions across different 7 domains: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal (mixed upper and diarrhea), constipation, bladder, and pupillomotor function. Single cumulative weighted score designed to reflect global autonomic dysfunction. Score is 0-100, greater than or = to 20 suggests moderate to severe autonomic dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kaplan, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai West, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No